CLINICAL TRIAL: NCT00005093
Title: A Randomized Double-Blind, Placebo-Controlled, Multicenter Study of CI-994 Capsules Plus Gemcitabine Infusion Versus Placebo Capsules Plus Gemcitabine Infusion as Second-Line Treatment of Patients With Advanced Nonsmall Cell Lung Cancer
Brief Title: Gemcitabine With or Without CI-994 in Treating Patients With Advanced Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: PD-994-013; CDR0000067735; ILEX-994-013
Record Dates: First submitted 2000-04-06; First posted 2004-06-18 (Estimated); Last update posted 2012-08-10 (Estimated); Status verified 2012-08

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Gemcitabine; tacedinaline

INTERVENTIONS:
Drug: gemcitabine hydrochloride
Drug: tacedinaline

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known whether gemcitabine plus CI-994 is more effective than gemcitabine alone for non-small cell lung cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of gemcitabine with or without CI-994 in treating patients who have advanced non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the efficacy and safety of gemcitabine with or without CI-994 in patients with advanced non-small cell lung cancer.

OUTLINE: This is a randomized, double blind, placebo controlled, multicenter study. Patients are stratified according to performance status and are randomized to one of two treatment arms. Arm I: Patients receive CI-994 orally on days 1-21 and gemcitabine IV over 30 minutes on days 1, 8, and 15. Arm II: Patients receive placebo capsules orally on days 1-21 and gemcitabine as in arm I. Treatment repeats every 28 days as long as medically appropriate (absence of disease progression or unacceptable toxicity).

PROJECTED ACCRUAL: A total of 176 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed recurrent, locally advanced, or metastatic, unresectable non-small cell lung cancer Failed or relapsed after one prior platinum containing regimen (cisplatin or carboplatin) as first line therapy Prior brain metastases allowed if resection and/or radiotherapy completed, no worsening of CNS symptoms, and at least 1 month since prior corticosteroids

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 70-100% Life expectancy: Greater than 12 weeks Hematopoietic: Absolute neutrophil count at least 2,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) AST or ALT no greater than 3 times ULN (no greater than 5 times ULN in patients with liver metastases) Renal: Creatinine clearance at least 50 mL/min Other: Able to swallow intact study capsules No active infection No life threatening illness (other than tumor) No prior malignancy within the past 5 years except well controlled nonmelanomatous skin cancer Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics At least 4 weeks since prior chemotherapy No more than one prior regimen of chemotherapy No prior gemcitabine No prior CI-994 At least 4 weeks since prior maintenance or consolidation therapy (e.g., matrix metalloprotein inhibitors) Endocrine therapy: See Disease Characteristics Radiotherapy: See Disease Characteristics At least 4 weeks since prior radiotherapy to primary site Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-12; Study Completion 2001-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Kimmel, PhD, Study Chair — Pfizer Incorporated - Ann Arbor
Locations (16):
- United States (9):
  - Cedars-Sinai Comprehensive Cancer Center, Los Angeles, California
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - New England Medical Center Hospital, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Raleigh Hematology/Oncology Associates - Wake Practice, Raleigh, North Carolina
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - West Clinic, P.C., Memphis, Tennessee
  - Southwest Regional Cancer Center, Austin, Texas
- Canada (7):
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Cancer Agency - Fraser Valley Cancer Centre, Surrey, British Columbia
  - BC Cancer Agency, Vancouver, British Columbia
  - British Columbia Cancer Agency - Vancouver Island Cancer Centre, Victoria, British Columbia
  - Ottawa Regional Cancer Center - General Division, Ottawa, Ontario
  - Mount Sinai Hospital - Toronto, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario